CLINICAL TRIAL: NCT01270269
Title: ACT-ICU Study: Activity and Cognitive Therapy in the Intensive Care Unit
Acronym: ACT-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Nathan Brummel, Assistant Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101037
Record Dates: First submitted 2010-11-02; First posted 2011-01-05 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Brain Injuries; Dementia; Myopathies; Muscle Disorders
Keywords: Asthenia; Muscle Weakness; Brain Injuries; Critical Illness; Critical Illness Myoneuropathy; Rehabilitation; Sepsis; Respiratory Failure; Delirium; Over-sedation; Immobility; Aging; Signs and Symptoms; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Manifestations; Neurologic Manifestations; Pathologic Processes; Brain Diseases; Central Nervous System Diseases; Craniocerebral Trauma; Trauma, Nervous System; Wounds and Injuries; Disorders of Environmental Origin
MeSH Terms: conditions — Brain Injuries; Dementia; Muscular Diseases; Asthenia; Muscle Weakness; Critical Illness; Sepsis; Respiratory Insufficiency; Delirium; Signs and Symptoms; Musculoskeletal Diseases; Neuromuscular Manifestations; Neurologic Manifestations; Pathologic Processes; Brain Diseases; Central Nervous System Diseases; Craniocerebral Trauma; Trauma, Nervous System; Wounds and Injuries; Disorders of Environmental Origin | interventions — Cognitive Training; Restraint, Physical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients (Controls) (No Intervention): Patients (Controls) will not receive formal (study-related) rehabilitation interventions and will only receive usual care.
- Behavioral: Phys & Func Rehab (Experimental): A multi-component program of physical rehabilitation interventions (without cognitive rehabilitation) will be delivered to patients beginning in the ICU and continue throughout the hospitalization.
  Interventions: Behavioral: Behavioral: Physical and functional rehabilitation
- Behavioral: Cog/Phys/Func Rehab (Experimental): A multi-component program of cognitive, physical, and functional rehabilitation interventions will be delivered to patients beginning in the ICU with continued cognitive rehabilitation in their home environments over a focused 12-week period.
  Interventions: Behavioral: Behavioral: Cognitive, physical, & functional rehabilitation

INTERVENTIONS:
Behavioral: Behavioral: Physical and functional rehabilitation — A multi-component program of physical rehabilitation interventions (without cognitive rehabilitation) will be delivered to patients beginning in the ICU and continue throughout the hospitalization.
  Other Names: cognitive rehabilitation
  Arms: Behavioral: Phys & Func Rehab
Behavioral: Behavioral: Cognitive, physical, & functional rehabilitation — A multi-component program of cognitive, physical, and functional rehabilitation interventions will be delivered to patients beginning in the ICU with continued cognitive rehabilitation in their home environments over a focused 12-week period.
  Other Names: cognitive rehabilitation
  Arms: Behavioral: Cog/Phys/Func Rehab

SUMMARY:
Intensive care unit (ICU) hospitalization saves lives but often does so at a high personal cost to ICU survivors who frequently experience significant cognitive impairment and an array of physical and functional disabilities that limit their recovery and quality of life. While the problems experienced by these patients are likely amenable to rehabilitation, few ICU survivors receive focused rehabilitation. Recently, early physical rehabilitation in ICU patients has shown to improve the chances a patient will regain their pre-hospital functional status. Early cognitive rehabilitation for these patients has not yet been explored. This pilot study will determine the feasibility of early cognitive rehabilitation in ICU patients. The investigators will perform cognitive and physical rehabilitation, beginning in the earliest phases of critical illness, to determine the effect of these therapies on cognitive and functional outcomes in ICU survivors. The investigators hypothesize that combined cognitive and physical rehabilitation, started in the ICU, will improve recovery of cognitive and physical function as well as improve quality of life of ICU survivors.

DETAILED DESCRIPTION:
The long-term consequences of critical illness and intensive care unit (ICU) hospitalization in ICU survivors are profound and include cognitive, physical, and functional impairments. The purpose of this study is to pilot test a multi-component, cognitive and physical rehabilitation program beginning in the ICU, combined with a 12-week home-based cognitive rehabilitation program following hospital discharge to determine whether participation in a rehabilitation program will result in improved outcomes among ICU survivors. The study will rely on a randomized controlled clinical trial design, with patients assigned to one of three groups: a "usual care" control group, an early physical activity group (without cognitive therapy), or an early cognitive therapy and physical activity group. All individuals in the intervention groups will receive protocolized physical therapy while hospitalized. In addition, individuals in the early cognitive therapy and physical activity group will receive cognitive therapy starting in the ICU and continuing for 12 weeks once a patient leaves the hospital. In-home visits will occur every other week during the 12-week intervention period.

The study's primary outcome is executive functioning (e.g. ability to plan, organize, multi-task) at 3-months following hospital discharge as measured by the Tower Test, a psychometric tool evaluating executive abilities. This has been chosen due to the fact that available research points to the presence of significant deficits in executive functioning among ICU survivors. Secondary outcomes include global cognitive function, physical function and Health Related Quality of Life by assessing scores on the following measures: Katz's ADL, Functional Activities Questionnaire, AD8, Short-Informant Questionnaire of Cognitive Decline in the Elderly, Clinical Dementia Rating Scale (if performed), Timed Up & Go test, Mini-Mental State Exam, Dysexecutive Questionnaire, Activities-Specific Balance Confidence Scale, Behavior Rating Inventory of Executive Function, Behavior Pain Inventory, Trails A & B test, Repeatable Battery for Assessment of Neuropsychological Status, General Employment Questionnaire, Beck Depression Inventory II, Post-traumatic stress checklist, Short Form 36, Canadian Study of Health and Aging and patient weight, and Tower Test score at 12 month follow-up. We will also track readmission to the hospital and admission to a nursing home or skilled rehabilitation facility as secondary outcomes during the 12-month follow-up period. The study duration will include 1 year of enrollment and 1 year for study completion following enrollment of the final patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the medical or surgical ICU who are receiving treatment for respiratory failure, cardiogenic shock, hemorrhagic shock, and/or septic shock.

Exclusion Criteria:

* Moderate to severe dementia on ICU admission based on a standardized surrogate assessment (as this would prohibit patients from functioning independently at home);
* Moderate or severe physical dysfunction that precludes performance of independent activities of daily living based on a standardized surrogate assessment;
* Live greater than 120 miles from Nashville;
* Blind, deaf, or unable to speak English;
* Prisoners;
* Homelessness and no secondary contact person available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Tower Test | 3 months post hospital discharge
  A psychometric measure of executive functioning.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) | 3 months post hospital discharge
  A timed test assessing physical strength and gait speed.
Functional Activities Questionnaire | 3 months post hospital discharge
  A brief measure of higher order (IADL) functioning.
EQ-5 Global Scores | 3 months post hospital discharge
  The EQ-5 Global Scores is an assessment of quality of life.
Katz Activities of Daily Living (ADL) scale | 3 months post hospital discharge
  A six-item tool assessing the degree of independence vs. dependence in basic activities of daily living.
Activities-Specific Balance Confidence Scale (ABC) | 3 months post hospital discharge
  A brief rating scale that asks participants to rate how confident they are that they can maintain their balance and remain steady while engaged in 16 non-hazardous tasks.
AD8 | 3 months post hospital discharge
  A brief surrogate or patient based measure that assesses recent change in a variety of cognitive abilities.
Short-Informant Questionnaire of Cognitive Decline in the Elderly (Short IQCODE) | 3 months post hospital discharge
  A measure of cognitive functioning that evaluates the degree of decline from baseline and which is complementary to the AD8. This measure will only be used in patients over the age of 50 who had any problems with memory or thinking prior to current illness.
Mini Mental State Exam (MMSE) | 3 months post hospital discharge
  A widely used measure of overall cognitive functioning that briefly samples abilities in a wide array of areas including memory and attention.
Dysexecutive Questionnaire (Dys Exec) | 3 months post hospital discharge
  A questionnaire, which has both patient and surrogate versions, that assesses patient functioning in a number of functional areas sensitive to executive dysfunction.
TRAILS A & B Test | 3 months post hospital discharge
  Two widely used to test the speed that it takes to connect a series of numbers (Part A) and numbers alternating with letters (Part B).
General and Employment Questionnaire | 3 months post hospital discharge
  A brief series of questions which pertain to patient history and demographics and which also inquire about employment both before and after ICU hospitalization.
Canadian Study of Health and Aging (CHSA) Frailty Scale | 3 months post hospital discharge
  A brief global rating scale of frailty based on clinical impression.
Tower Test | 12 months post hospital discharge
  A psychometric measure of executive functioning.
Timed Up and Go (TUG) | 12 months post hospital discharge
  A timed test assessing physical strength and gait speed.
Functional Activities Questionnaire | 12 months post-hospital discharge
  A brief measure of higher order (IADL) functioning.
EQ-5 Global Scores | 12 months post hospital discharge
  The EQ-5 Global Scores is an assessment of quality of life.
Katz Activities of Daily Living (ADL) scale | 12 months post hospital discharge
  A six-item tool assessing the degree of independence vs. dependence in basic activities of daily living.
Activities-Specific Balance Confidence Scale (ABC) | 12 months post hospital discharge
  A brief rating scale that asks participants to rate how confident they are that they can maintain their balance and remain steady while engaged in 16 non-hazardous tasks.
AD8 | 12 months post hospital discharge
  A brief surrogate or patient based measure that assesses recent change in a variety of cognitive abilities.
Short-Informant Questionnaire of Cognitive Decline in the Elderly (Short IQCODE) | 12 months post hospital discharge
  A measure of cognitive functioning that evaluates the degree of decline from baseline and which is complementary to the AD8. This measure will only be used in patients over the age of 50 who had any problems with memory or thinking prior to current illness.
Mini Mental State Exam (MMSE) | 12 months post hospital discharge
  A widely used measure of overall cognitive functioning that briefly samples abilities in a wide array of areas including memory and attention.
Dysexecutive Questionnaire (Dys Exec) | 12 months post hospital discharge
  A questionnaire, which has both patient and surrogate versions, that assesses patient functioning in a number of functional areas sensitive to executive dysfunction.
TRAILS A & B Test | 12 months post hospital discharge
  Two widely used to test the speed that it takes to connect a series of numbers (Part A) and numbers alternating with letters (Part B).
General and Employment Questionnaire | 12 months post hospital discharge
  A brief series of questions which pertain to patient history and demographics and which also inquire about employment both before and after ICU hospitalization.
Canadian Study of Health and Aging (CHSA) Frailty Scale | 12 months post hospital discharge
  A brief global rating scale of frailty based on clinical impression.
Mortality | 2 months post hospital discharge
Rehospitalization rate and number of hospital days | 12 months post hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Nathan E. Brummel, MD, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Schweickert WD, Herlitz J, Pohlman AS, Gehlbach BK, Hall JB, Kress JP. A randomized, controlled trial evaluating postinsertion neck ultrasound in peripherally inserted central catheter procedures. Crit Care Med. 2009 Apr;37(4):1217-21. doi: 10.1097/CCM.0b013e31819cee7f. PMID 19242336
- [Background] Brummel NE, Jackson JC, Girard TD, Pandharipande PP, Schiro E, Work B, Pun BT, Boehm L, Gill TM, Ely EW. A combined early cognitive and physical rehabilitation program for people who are critically ill: the activity and cognitive therapy in the intensive care unit (ACT-ICU) trial. Phys Ther. 2012 Dec;92(12):1580-92. doi: 10.2522/ptj.20110414. Epub 2012 May 10. PMID 22577067
- [Background] Jackson JC, Ely EW, Morey MC, Anderson VM, Denne LB, Clune J, Siebert CS, Archer KR, Torres R, Janz D, Schiro E, Jones J, Shintani AK, Levine B, Pun BT, Thompson J, Brummel NE, Hoenig H. Cognitive and physical rehabilitation of intensive care unit survivors: results of the RETURN randomized controlled pilot investigation. Crit Care Med. 2012 Apr;40(4):1088-97. doi: 10.1097/CCM.0b013e3182373115. PMID 22080631
- [Result] Brummel NE, Girard TD, Ely EW, Pandharipande PP, Morandi A, Hughes CG, Graves AJ, Shintani A, Murphy E, Work B, Pun BT, Boehm L, Gill TM, Dittus RS, Jackson JC. Feasibility and safety of early combined cognitive and physical therapy for critically ill medical and surgical patients: the Activity and Cognitive Therapy in ICU (ACT-ICU) trial. Intensive Care Med. 2014 Mar;40(3):370-9. doi: 10.1007/s00134-013-3136-0. Epub 2013 Nov 21. PMID 24257969